CLINICAL TRIAL: NCT06864663
Title: A Comparative Study of Combined Ultrasound-Guided Adductor Canal Block and Interspace Between the Popliteal Artery and Capsule of the Knee (IPACK) Versus Combined Adductor Canal Block and Genicular Nerve Block Following Total Knee Arthroplasty
Brief Title: A Comparative Study of Combined Adductor Canal and Interspace Between Popliteal Artery and Knee Capsule Versus Combined Adductor Canal and Genicular Nerve in Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R313/2024
Record Dates: First submitted 2025-02-21; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-01

CONDITIONS: Nerve Block; Regional Anaesthesia
Keywords: adductor canal block; interspace between popliteal artery and capsule of knee; knee arthroplasty; genicular nerve block
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Intervention Model Description: Randomized controlled interventional prospective study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving combined ACB and IPACK blocks (Active Comparator): ultrasound guided block of saphenous nerve in adductor canal and block of articular branches of knee between the popliteal artery and the knee capsule (IPACK)
  Interventions: Drug: Nerve Block with bupivacaine 0.25%
- Patients receiving combined ACB and GNB (Active Comparator): ultrasound guided block of saphenous nerve in adductor canal and block of the three peri-knee nerve branches: the superior medial genicular nerve (SMGN), inferior medial genicular nerve (IMGN), and superior lateral genicular nerve (SLGN)
  Interventions: Drug: nerve block with bupivacaine 0.25%

INTERVENTIONS:
Drug: nerve block with bupivacaine 0.25% — ultrasound guided adductor canal block and interspace between the popliteal artery and the knee capsule using bupivacaine 0.25%
  Arms: Patients receiving combined ACB and GNB
Drug: Nerve Block with bupivacaine 0.25% — ultrasound guided combined adductor canal block and genicular nerve block using bupivacaine 0.25%
  Arms: Patients receiving combined ACB and IPACK blocks

SUMMARY:
The aim of this study is to investigate the effectiveness of combined adductor canal block (ACB) with interspace between popliteal artery and the knee capsule (IPACK) versus combined ACB with genicular nerve block (GNB) for providing analgesia in knee arthroplasty. The investigators hypothesize that the analgesic efficacy of ACB combined with GNB will be non-inferior to that of ACB combined with IPACK. Additionally, the investigators aim to assess whether the combination of ACB and GNB results in a significantly lower occurrence of sensory or motor block affecting the tibial and common peroneal nerves compared to ACB and IPACK

DETAILED DESCRIPTION:
Spinal anesthesia will be chosen as the main anesthetic technique by injecting 3-3.5 ml of hyperbaric bupivacaine 0.5% by 24 G pencil-point needle at lumbar (L2-L3) or (L3-L4) space with 25 ug of fentanyl as adjuvant while patient is in setting position.

In both groups, the adductor canal block (ACB) will be performed with the patient in a supine position, the operative limb externally rotated, and the knee slightly flexed. A high-frequency ultrasound probe (10-15 MHz) will be positioned at the mid-thigh, at the midpoint of the line connecting the patella to the anterior superior iliac spine.

During the procedure, the following structures will be identified: the femoral artery, femoral vein, sartorius muscle, vastus medialis, and adductor longus. The hyperechoic appearance of the saphenous nerve will be visualized lateral to the femoral artery. Using an in-plane technique, 15 mL of 0.25% bupivacaine will be injected to achieve effective analgesia.

For (Group A) To perform the interspace between popliteal artery and knee capsule (IPACK) block, a curvilinear ultrasound probe (2-5 MHz) will first be positioned on the lower third of the medial thigh to identify the femoral vessels. The transducer will then be moved caudally into the popliteal fossa, allowing visualization of the femoral artery as it transitions into the popliteal artery. With the knee flexed at 90°, the needle will be advanced using an in-plane ultrasound-guided technique. The needle trajectory will be from medial to lateral, targeting the space between the popliteal vessels and the posterior capsule of the knee joint. Once the needle tip is positioned approximately 2 cm beyond the lateral border of the popliteal artery, an injection of 15 mL of 0.25% bupivacaine will be administered into this interspace.

For (Group B), The genicular nerve block (GNB) will target three peri-knee nerve branches: the superior medial genicular nerve (SMGN), inferior medial genicular nerve (IMGN), and superior lateral genicular nerve (SLGN). Each nerve will receive an injection of 5 mL of 0.25% bupivacaine.

For SMGN block the high frequency ultrasound probe will be placed laterally over the medial supracondylar area of the femur to identify the SMGN near the superior medial genicular artery, followed by injection adjacent to the artery. For the IMGN, the probe will be positioned over the medial condyle of the tibia to locate the inferior medial genicular artery near the neck of the tibia, again injecting adjacent to the artery. Finally, the SLGN will be targeted by placing the probe over the lateral condyle of the femur to find the superior lateral genicular artery, with the local anesthetic injected nearby.

The investigators will omit the inferolateral genicular nerve (ILGN) block to prevent any unwanted motor weakness or the potential for foot drop that may occur from inadvertently blocking branches of the common peroneal nerve. This decision aligns with the goal of optimizing analgesia while minimizing the risk of motor deficits, ensuring a safer and more effective postoperative recovery for patients undergoing knee arthroplasty.

In postoperative period all patients will receive the same adjuvant multimodal analgesia which will be 1000 mg of paracetamol with or without 30 mg ketorolac depending on comorbidities

ELIGIBILITY:
Inclusion Criteria:

1. Patients American Society of anesthesiologists' physical status (ASA) I to III.
2. Aged 18 to 70 years.
3. Both sexes.
4. Patients scheduled for total knee arthroplasty.

Exclusion Criteria:

1. Patient refusal
2. ASA physical status IV or more.
3. Patients with known allergy to any of the study drugs.
4. Infection at the site of injection.
5. Patients with neuromuscular disease.
6. Presence of any coagulopathy.
7. Patients with history of any psychiatric or cognitive disorder.
8. patient with previous knee surgery.
9. BMI more than 40 kg/m2.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
individual visual analog pain scores at 0, 6, 12 , 24 and 48 h postoperatively | 48 hours
  (VAS; 0 = no pain and 10 = worst pain imaginable)

SECONDARY OUTCOMES:
time to first reported pain and first analgesic request during post-anesthesia care unit stay | 48 hours
  reported time in minutes
Analgesic consumption during the first 48 h post-surgery | 48 hours
  Converted to IV pethidine equivalents. The analgesic dose of pethidine will be 0.5 mg/kg/dose to be repeated on demand
Quadriceps muscle strength | 24 hours
  will be measured using the Straight Leg Raise (SLR) test, which will be conducted preoperatively and again 24 hours postoperatively. The SLR will be scored on a scale from 0 to 5, where 0 indicates no voluntary contraction, 1 signifies muscle flicker without limb movement, 2 represents active movement with gravity eliminated, 3 indicates movement against gravity but without resistance, 4 denotes movement against some resistance, and 5 reflects normal motor strength against resistance.
The sensorimotor functions of the tibial nerve and common peroneal nerve (CPN) will be evaluated using a 3-point scale | 8 hours postoperative
  For sensory function, the scale will be as follows: 0 indicates normal sensation, 1 signifies lack of cold perception but intact touch sensation, and 2 denotes absence of touch sensation. For motor function, the scale will be: 0 for normal motor function, 1 for deficient motor function, and 2 for no motor function.
Ambulation and mobilization ability | 48 hours
  Assessed using the Timed Up and Go (TUG) test

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: from 20/2/2025 to 20/9/2025
Access Criteria: All researchers

REFERENCES:
- [Background] Kukreja P, Venter A, Mason L, Kofskey AM, Northern T, Naranje S, Ghanem E, Lawson PA, Kalagara H. Comparison of Genicular Nerve Block in Combination With Adductor Canal Block in Both Primary and Revision Total Knee Arthroplasty: A Retrospective Case Series. Cureus. 2021 Jul 29;13(7):e16712. doi: 10.7759/cureus.16712. eCollection 2021 Jul. PMID 34471571
- [Background] Padhy S, Patki AY, Kar AK, Durga P, Sireesha L. Comparison of sensory posterior articular nerves of the knee (SPANK) block versus infiltration between the popliteal artery and the capsule of the knee (IPACK) block when added to adductor canal block for pain control and knee rehabilitation after total knee arthroplasty---A prospective randomised trial. Indian J Anaesth. 2021 Nov;65(11):792-797. doi: 10.4103/ija.ija_682_21. Epub 2021 Nov 23. PMID 35001951
- [Background] Gonzalez Sotelo V, Macule F, Minguell J, Berge R, Franco C, Sala-Blanch X. Ultrasound-guided genicular nerve block for pain control after total knee replacement: Preliminary case series and technical note. Rev Esp Anestesiol Reanim. 2017 Dec;64(10):568-576. doi: 10.1016/j.redar.2017.04.001. Epub 2017 May 26. English, Spanish. PMID 28554709
- [Background] Mu T, Yuan B, Wei K, Yang Q. Adductor canal block combined with genicular nerve block versus local infiltration analgesia for total knee arthroplasty: a randomized noninferiority trial. J Orthop Surg Res. 2024 Sep 6;19(1):546. doi: 10.1186/s13018-024-05048-5. PMID 39238029
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36931354/